CLINICAL TRIAL: NCT06794892
Title: Comparative Outcomes of One-Anastomosis Gastric Bypass and Roux-en-Y Gastric Bypass As Revisional Procedures Following Failed Restrictive Bariatric Surgery: a Prospective Multicenter Study with Three-Year Follow-Up
Brief Title: Comparative Outcomes of One-Anastomosis Gastric Bypass and Roux-en-Y Gastric Bypass As Revisional Procedures Following Failed Restrictive Bariatric Surgery
Acronym: COBRA stady
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Principal Investigator, PhD. MD,, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 2025010188
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Obesity, Morbid; Type 2 Diabetes Mellitus (T2DM); Hypertension; Dyslipidemia
Keywords: obesity; One anastomosis gastric bypass; Roux and Y gastric Bypass
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OAGB Cohort - Patients undergoing One-Anastomosis Gastric Bypass as a revisional procedure.: OAGB Cohort: This group consists of patients who underwent One-Anastomosis Gastric Bypass (OAGB) as a revisional bariatric procedure following insufficient weight loss or weight regain after primary restrictive surgeries, such as laparoscopic sleeve gastrectomy (LSG) or laparoscopic adjustable gastric banding (LAGB). These patients were monitored over three years to evaluate outcomes, including weight loss, complication rates, and improvement in obesity-related comorbidities.
- RYGB Cohort - Patients undergoing Roux-en-Y Gastric Bypass as a revisional procedure.: RYGB Cohort: This group includes patients who underwent Roux-en-Y Gastric Bypass (RYGB) as a revisional bariatric procedure due to insufficient weight loss or significant weight regain after primary restrictive surgeries, such as laparoscopic sleeve gastrectomy (LSG) or laparoscopic adjustable gastric banding (LAGB). The cohort was followed prospectively over three years to assess outcomes, including weight loss, resolution of obesity-related comorbidities, complication rates, and overall surgical success.

SUMMARY:
Study Description

This prospective, multicenter study aims to compare the outcomes of One-Anastomosis Gastric Bypass (OAGB) and Roux-en-Y Gastric Bypass (RYGB) as revisional procedures for patients experiencing insufficient weight loss or weight regain following restrictive bariatric surgeries, such as laparoscopic sleeve gastrectomy (LSG) or laparoscopic adjustable gastric banding (LAGB). Conducted between January 2019 and December 2021, the study involves a three-year follow-up of 328 patients across high-volume bariatric centers.

The primary objective is to evaluate the effectiveness of these revisional procedures in achieving additional weight loss. Secondary objectives include analyzing differences in operative times, complication rates (short- and long-term), reduction of obesity-related comorbidities, mortality, and overall patient outcomes.

This study uniquely integrates comprehensive pre- and postoperative assessments, including radiological evaluations, to better understand predictors of success and provide evidence for optimal surgical strategies in revisional bariatric care.

DETAILED DESCRIPTION:
Study Objective and Design

The primary objective of this multicenter study was to compare the effectiveness of one-anastomosis gastric bypass and Roux-en-Y gastric bypass as revisional procedures for addressing insufficient weight loss or weight regain following failed primary restrictive bariatric surgery. Effectiveness was measured in terms of additional weight loss. Secondary objectives included comparisons of surgical duration, reduction in obesity-related comorbidities, rates of short- and long-term complications, and mortality between the two revisional approaches. The study was conducted from January 2019 to December 2021, with a three-year follow-up for each participant.

Patient Selection and Data Collection

Participants were recruited from four high-volume bariatric centers in Italy. Inclusion criteria encompassed adults aged 18 to 65 years who exhibited insufficient weight loss, defined as excess weight loss of less than 50%, total weight loss of less than 25%, or a BMI greater than 40 kg/m² at least two years after undergoing laparoscopic sleeve gastrectomy or laparoscopic adjustable gastric banding. Eligible patients were those requiring revisional surgery exclusively for inadequate weight loss or regain. Exclusion criteria included revisional surgery for other indications (e.g., complications such as stenosis or severe gastroesophageal reflux), untreated psychiatric illness, active eating disorders, pregnancy, or any previous gastric surgery unrelated to bariatric interventions.

Preoperative assessments involved a multidisciplinary team including an endocrinologist, dietitian, and psychologist. Patients identified with maladaptive eating patterns received treatment before surgery to optimize outcomes. Baseline data on demographics, preoperative BMI, and comorbidities were collected and followed up throughout the study. Ethical approval was obtained from all participating centers' medical ethics committees.

Surgical Technique and Perioperative Management

One-Anastomosis Gastric Bypass

The surgical protocol for one-anastomosis gastric bypass involved removing the gastric band in patients previously treated with laparoscopic adjustable gastric banding, followed by dissection of the angle of His. If present, the fibrous capsule from the band was excised. A gastric pouch was created by horizontally transecting the stomach at the junction of the corpus and antrum, typically at the level of the crow's foot. For patients with a prior sleeve gastrectomy, the residual sleeve was horizontally transected. The length of the biliopancreatic limb was tailored based on the patient's preoperative BMI, ranging from 180 to 200 cm.

Roux-en-Y Gastric Bypass

For Roux-en-Y gastric bypass, the gastric band and fibrous capsule were removed in previously banded patients, followed by adhesiolysis as necessary. A small gastric pouch was created by transecting the stomach. The lengths of the alimentary and biliopancreatic limbs were standardized across centers. Closure of mesenteric defects was performed at the surgeon's discretion.

Data Collection

Type 2 Diabetes Mellitus

Type 2 diabetes mellitus was diagnosed according to established guidelines, based on fasting plasma glucose readings above 126 mg/dL, a two-hour glucose level exceeding 200 mg/dL during an oral glucose tolerance test, or a glycated hemoglobin level above 6.5%. Complete remission was defined as fasting plasma glucose levels below 100 mg/dL and HbA1c less than 6.0% without antidiabetic medications. Follow-ups were conducted at 3, 6, 12, 24, and 36 months post-revision.

Hypertension

Hypertension was defined as systolic blood pressure greater than or equal to 140 mmHg or diastolic pressure greater than or equal to 90 mmHg. Remission was defined as achieving blood pressure below 120/80 mmHg without antihypertensive medications. Blood pressure measurements were taken at 3, 6, 12, 24, and 36 months.

Obstructive Sleep Apnea Syndrome

Obstructive sleep apnea was diagnosed based on prior polysomnography, with an Apnea-Hypopnea Index exceeding 15 events/hour or more than 5 events/hour in the presence of related symptoms such as snoring or daytime sleepiness. Remission was defined by resolution of these symptoms. Follow-up assessments occurred at 3, 6, 12, 24, and 36 months.

Outcome Measures

Baseline characteristics, including demographics, preoperative BMI, and comorbidities, were recorded at study entry.

Primary Outcomes

* Percentage Total Weight Loss: Measured as the proportion of total body weight lost relative to initial weight.
* Percentage Excess BMI Loss: Calculated as the proportion of BMI lost relative to the amount exceeding a BMI of 25.

Secondary Outcomes

* Mortality: Measured throughout the three-year follow-up.
* Complications: Assessed using the Clavien-Dindo classification. Short-term complications included anastomotic leaks, bleeding, infections, perforations, myocardial infarction, and stroke. Long-term complications included nutritional deficiencies, gastric ulcers, strictures, bile reflux, internal herniation, and malnutrition.
* Comorbidity Improvement: Evaluated using standardized criteria for resolution or improvement of type 2 diabetes, cardiovascular disease, obstructive sleep apnea, dyslipidemia, and osteoarthritis.

Quality of Life Outcomes

Quality of life was assessed using validated tools such as the SF-36 at multiple intervals: baseline, and 3, 6, 12, 24, and 36 months post-surgery. Domains evaluated included physical health, mobility, social functioning, emotional well-being, and fatigue. Quality-of-life trends were compared between the two surgical groups to identify differences in patient-reported outcomes.

This structured approach provides a comprehensive evaluation of surgical and patient-centered outcomes in revisional bariatric surgery.Study Objective and Design

The primary objective of this multicenter study was to compare the effectiveness of one-anastomosis gastric bypass and Roux-en-Y gastric bypass as revisional procedures for addressing insufficient weight loss or weight regain following failed primary restrictive bariatric surgery. Effectiveness was measured in terms of additional weight loss. Secondary objectives included comparisons of surgical duration, reduction in obesity-related comorbidities, rates of short- and long-term complications, and mortality between the two revisional approaches. The study was conducted from January 2019 to December 2021, with a three-year follow-up for each participant.

Patient Selection and Data Collection

Participants were recruited from four high-volume bariatric centers in Italy. Inclusion criteria encompassed adults aged 18 to 65 years who exhibited insufficient weight loss, defined as excess weight loss of less than 50%, total weight loss of less than 25%, or a BMI greater than 40 kg/m² at least two years after undergoing laparoscopic sleeve gastrectomy or laparoscopic adjustable gastric banding. Eligible patients were those requiring revisional surgery exclusively for inadequate weight loss or regain. Exclusion criteria included revisional surgery for other indications (e.g., complications such as stenosis or severe gastroesophageal reflux), untreated psychiatric illness, active eating disorders, pregnancy, or any previous gastric surgery unrelated to bariatric interventions.

Preoperative assessments involved a multidisciplinary team including an endocrinologist, dietitian, and psychologist. Patients identified with maladaptive eating patterns received treatment before surgery to optimize outcomes. Baseline data on demographics, preoperative BMI, and comorbidities were collected and followed up throughout the study. Ethical approval was obtained from all participating centers' medical ethics committees.

Surgical Technique and Perioperative Management

One-Anastomosis Gastric Bypass

The surgical protocol for one-anastomosis gastric bypass involved removing the gastric band in patients previously treated with laparoscopic adjustable gastric banding, followed by dissection of the angle of His. If present, the fibrous capsule from the band was excised. A gastric pouch was created by horizontally transecting the stomach at the junction of the corpus and antrum, typically at the level of the crow's foot. For patients with a prior sleeve gastrectomy, the residual sleeve was horizontally transected. The length of the biliopancreatic limb was tailored based on the patient's preoperative BMI, ranging from 180 to 200 cm.

Roux-en-Y Gastric Bypass

For Roux-en-Y gastric bypass, the gastric band and fibrous capsule were removed in previously banded patients, followed by adhesiolysis as necessary. A small gastric pouch was created by transecting the stomach. The lengths of the alimentary and biliopancreatic limbs were standardized across centers. Closure of mesenteric defects was performed at the surgeon's discretion.

Data Collection

Type 2 Diabetes Mellitus

Type 2 diabetes mellitus was diagnosed according to established guidelines, based on fasting plasma glucose readings above 126 mg/dL, a two-hour glucose level exceeding 200 mg/dL during an oral glucose tolerance test, or a glycated hemoglobin level above 6.5%. Complete remission was defined as fasting plasma glucose levels below 100 mg/dL and HbA1c less than 6.0% without antidiabetic medications. Follow-ups were conducted at 3, 6, 12, 24, and 36 months post-revision.

Hypertension

Hypertension was defined as systolic blood pressure greater than or equal to 140 mmHg or diastolic pressure greater than or equal to 90 mmHg. Remission was defined as achieving blood pressure below 120/80 mmHg without antihypertensive medications. Blood pressure measurements were taken at 3, 6, 12, 24, and 36 months.

Obstructive Sleep Apnea Syndrome

Obstructive sleep apnea was diagnosed based on prior polysomnography, with an Apnea-Hypopnea Index exceeding 15 events/hour or more than 5 events/hour in the presence of related symptoms such as snoring or daytime sleepiness. Remission was defined by resolution of these symptoms. Follow-up assessments occurred at 3, 6, 12, 24, and 36 months.

Outcome Measures

Baseline characteristics, including demographics, preoperative BMI, and comorbidities, were recorded at study entry.

Primary Outcomes

* Percentage Total Weight Loss: Measured as the proportion of total body weight lost relative to initial weight.
* Percentage Excess BMI Loss: Calculated as the proportion of BMI lost relative to the amount exceeding a BMI of 25.

Secondary Outcomes

* Mortality: Measured throughout the three-year follow-up.
* Complications: Assessed using the Clavien-Dindo classification. Short-term complications included anastomotic leaks, bleeding, infections, perforations, myocardial infarction, and stroke. Long-term complications included nutritional deficiencies, gastric ulcers, strictures, bile reflux, internal herniation, and malnutrition.
* Comorbidity Improvement: Evaluated using standardized criteria for resolution or improvement of type 2 diabetes, cardiovascular disease, obstructive sleep apnea, dyslipidemia, and osteoarthritis.

Quality of Life Outcomes

Quality of life was assessed using validated tools such as the SF-36 at multiple intervals: baseline, and 3, 6, 12, 24, and 36 months post-surgery. Domains evaluated included physical health, mobility, social functioning, emotional well-being, and fatigue. Quality-of-life trends were compared between the two surgical groups to identify differences in patient-reported outcomes.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Adults aged 18-65 years.
* Experienced insufficient weight loss, defined as:
* Excess weight loss (EWL) < 50%.
* Total weight loss (TWL) < 25%.
* BMI > 40 kg/m² at least two years after primary restrictive surgery.
* Previously underwent laparoscopic sleeve gastrectomy (LSG) or laparoscopic adjustable gastric banding (LAGB).
* Undergoing revisional surgery specifically for inadequate weight loss or weight regain.

Exclusion Criteria:

* Revisional surgery performed for indications other than inadequate weight loss or weight regain (e.g., complications of the primary procedure such as stenosis or refractory gastroesophageal reflux, or for comorbidity management).
* Known psychiatric illness or untreated eating disorders.
* Pregnancy.
* History of prior gastric surgery unrelated to bariatric interventions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from a population of adults aged 18 to 65 years who have undergone primary restrictive bariatric surgery, such as laparoscopic sleeve gastrectomy (LSG) or laparoscopic adjustable gastric banding (LAGB), and have experienced insufficient weight loss or significant weight regain. This population will include individuals from multiple high-volume bariatric centers, ensuring a diverse cohort representing a range of demographic, clinical, and surgical characteristics.
  Eligible participants must meet specific criteria, such as a body mass index (BMI) ≤ 40 kg/m² and stable comorbid conditions. The study will focus on patients who require revisional bariatric surgery and are deemed suitable candidates for One-Anastomosis Gastric Bypass (OAGB) or Roux-en-Y Gastric Bypass (RYGB). Patients with specific contraindications, such as ongoing acute medical conditions or inability to provide informed consent, will be excluded to maintain the integrity and safety of
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage Total Weight Loss (%TWL) | Measured at 12 months post-surgery.
  The percentage of total body weight lost from the pre-revisional weight to the weight at 36 months post-revision.
Percentage Total Weight Loss (%TWL) | Measured at 24, months post-surgery.
  The percentage of total body weight lost from the pre-revisional weight to the weight at 36 months post-revision.
Percentage Total Weight Loss (%TWL) | Measured at 36 months post-surgery.
  The percentage of total body weight lost from the pre-revisional weight to the weight at 36 months post-revision.

SECONDARY OUTCOMES:
Percentage Excess BMI Loss (%EBMIL) | Measured at 12 months post-surgery
  The percentage reduction in excess BMI relative to an ideal BMI of 25, calculated at 12 months post-revision.
Percentage Excess BMI Loss (%EBMIL) | Measured at 24 months post-surgery
  The percentage change in excess BMI relative to an ideal BMI of 25, calculated at 24 months following revisional surgery. This measure evaluates the change in excess BMI to assess the effectiveness of the revisional bariatric procedure.
Percentage Excess BMI Loss (%EBMIL) | Measured at 36 months post-surgery
  The percentage change in excess BMI relative to an ideal BMI of 25, calculated at 24 months following revisional surgery. This measure evaluates the change in excess BMI to assess the effectiveness of the revisional bariatric procedure.
Reduction in Obesity-Related Comorbidities | 36 months
  Description: Improvement or resolution of comorbid conditions, including type 2 diabetes mellitus (T2DM), hypertension, dyslipidemia, and obstructive sleep apnea syndrome (OSAS).
Complication Rates | until 30 days follow-up period.
  Incidence of short-term (≤30 days) and long-term (>30 days) surgical complications, including anastomotic leaks, internal herniation, biliary reflux, and malnutrition.
Complication Rates | 36-month follow-up period.
  Incidence of short-term (≤30 days) and long-term (>30 days) surgical complications, including anastomotic leaks, internal herniation, biliary reflux, and malnutrition.
Mortality Rate | 36 months post-surgery.
  The percentage of patients who die from any cause during the 36-month follow-up period.
Quality of Life (QoL) Assessment | Baseline
  Description: Patient-reported outcomes measured using a validated tool such as the SF-36 or Bariatric Quality of Life Index
Quality of Life (QoL) Assessment | , 12 months post-surgery
  Description: Patient-reported outcomes measured using a validated tool such as the SF-36 or Bariatric Quality of Life Index
Quality of Life (QoL) Assessment | 24, months post-surgery months post-surgery
  Description: Patient-reported outcomes measured using a validated tool such as the SF-36 or Bariatric Quality of Life Index
Quality of Life (QoL) Assessment | 36 months post-surgery, months post-surgery months post-surgery
  Description: Patient-reported outcomes measured using a validated tool such as the SF-36 or Bariatric Quality of Life Index
Remission of Hypertension (HTN) | Measured at 3, months post-revision.
  Achieving normal blood pressure levels (< 120/80 mmHg) without the use of antihypertensive medications. Hypertension was defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
Remission of Hypertension (HTN) | Measured at 6, months post-revision.
  Achieving normal blood pressure levels (< 120/80 mmHg) without the use of antihypertensive medications. Hypertension was defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
Remission of Hypertension (HTN) | Measured at 12, months post-revision.
  Achieving normal blood pressure levels (< 120/80 mmHg) without the use of antihypertensive medications. Hypertension was defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
Remission of Hypertension (HTN) | Measured at 24, months post-revision.
  Achieving normal blood pressure levels (< 120/80 mmHg) without the use of antihypertensive medications. Hypertension was defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
Remission of Hypertension (HTN) | Measured at 36, months post-revision.
  Achieving normal blood pressure levels (< 120/80 mmHg) without the use of antihypertensive medications. Hypertension was defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
Type 2 Diabetes Mellitus (T2DM) | Assessed at 3,months post-revision
  Partial remission of Type 2 Diabetes Mellitus T2DM, defined as improved glycemic control with reduced medication doses but without meeting the criteria for complete remission.
Type 2 Diabetes Mellitus (T2DM) | Assessed at 6months post-revision
  Partial remission of Type 2 Diabetes Mellitus T2DM, defined as improved glycemic control with reduced medication doses but without meeting the criteria for complete remission.
Type 2 Diabetes Mellitus (T2DM) | Assessed at 12 months post-revision
  Partial remission of Type 2 Diabetes Mellitus T2DM, defined as improved glycemic control with reduced medication doses but without meeting the criteria for complete remission.
Type 2 Diabetes Mellitus (T2DM) | Assessed at 24 months post-revision
  Partial remission of Type 2 Diabetes Mellitus T2DM, defined as improved glycemic control with reduced medication doses but without meeting the criteria for complete remission.
Type 2 Diabetes Mellitus (T2DM) | Assessed at 36 months post-revision
  Partial remission of Type 2 Diabetes Mellitus T2DM, defined as improved glycemic control with reduced medication doses but without meeting the criteria for complete remission.

CONTACTS AND LOCATIONS:
Locations (1):
- Lacco Ameno Via Fundera 2, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: No